CLINICAL TRIAL: NCT00918463
Title: A Phase II, Single-Institution, Single-Arm, Open-Label Study to Evaluate the Safety and Efficacy of a Single Agent Dasatinib (Sprycel) in Subjects With Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Brief Title: A Study to Evaluate the Safety and Efficacy of Dasatinib (Sprycel) in Subjects With Relapsed or Refractory Diffuse Large B-Cell Lymphoma (DLBCL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early due to lack of accrual.
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0809009979
Record Dates: First submitted 2009-03-10; First posted 2009-06-11 (Estimated); Results first posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: lymphoma; diffuse; refractory
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- all patients (Experimental)
  Interventions: Drug: dasatinib

INTERVENTIONS:
Drug: dasatinib — 100 mg daily dosing
  Other Names: Sprycel

SUMMARY:
This is a Phase II, single institution, single-arm, open-label study of oral dasatinib monotherapy administered to subjects with relapsed or refractory aggressive DLBCL.

This study will be conducted in two phases: a Treatment Phase and a Follow-up Phase.

Research Hypothesis: Dasatinib, when administered orally at a continuous dose of 100 mg once daily, will be safe and effective in treating subjects that have failed prior therapies to diffuse large B cell lymphoma (DLBCL) or have relapsed disease.

ELIGIBILITY:
Inclusion Criteria:

* Must understand and voluntarily sign an informed consent form.
* Must be > = 18 years of age at the time of signing the informed consent form.
* Must be able to adhere to the study visit schedule and other protocol requirements.
* Biopsy-proven aggressive Diffuse Large B-Cell Lymphoma.
* Relapsed or refractory to previous therapy for lymphoma.
* Subjects must have received at least one prior combination chemotherapy regimen. There is no limit on the number of prior therapies.
* Subjects who have relapsed following an autologous stem cell transplant are eligible.
* Subjects must have measurable disease on cross sectional imaging that is at least 2 cm in the longest diameter.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2.
* Life expectancy of > = 90 days (3 months).
* Ability to take oral medication: dasatinib tablets may be swallowed as a whole.
* Adequate organ function:

Total bilirubin <2.0 times Upper Limit of Normal (ULN) Serum Na, K, Mg, Phos, and Ca > Lower Limit of Normal (LLN) Hemoglobin, neutrophil count, platelets, PT/PTT all grade 0-1 Serum creatinine concentration <1.5 x institutional upper limit of normal (ULN). Serum SGOT/AST or SGPT/ALT < 2.5 x institutional upper limit of normal (ULN).

* Concomitant medications:

  1. Patient agrees to discontinue St. Johns Wort while receiving dasatinib
  2. IV biphosphonates will be withheld for the first 8 weeks of dasatinib therapy due to risk of hypocalcemia.
* Females of childbearing potential (FCBP) must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse during the following time periods related to this study: 1) for at least 28 days before starting study drug; 2) while participating in the study; and 3) for at least 28 days after discontinuation from the study. The two methods of reliable contraception must include one highly effective method (i.e. intrauterine device (IUD), hormonal [birth control pills, injections, or implants], tubal ligation, partner's vasectomy) and one additional effective (barrier) method (i.e. latex condom, diaphragm, cervical cap). FCBP must be referred to a qualified provider of contraceptive methods if needed.
* Before starting study drug:
* Female Subjects: FCBP must have two negative pregnancy tests (sensitivity of at least 50 mIU/mL) prior to starting study drug. The first pregnancy test must be performed within 10-14 days prior to the start of study drug and the second pregnancy test must be performed within 24 hours prior to the start of study drug. The subject may not receive study drug until the Investigator has verified that the results of these pregnancy tests are negative; Will be warned that sharing study drug is prohibited and will be counseled about pregnancy precautions and potential risks of fetal exposure; Must agree to abstain from donating blood during study participation and for at least 28 days after discontinuation from the study.
* Male Subjects: Must agree to use a latex condom during sexual contact with females of childbearing potential while participating in the study and for at least 28 days following discontinuation from the study even if he has undergone a successful vasectomy; Will be warned that sharing study drug is prohibited and will be counseled about pregnancy precautions and potential risks of fetal exposure; Must agree to abstain from donating blood, semen, or sperm during study participation and for at least 28 days after discontinuation from the study.
* During study participation and for 28 days following discontinuation from the study:
* All Subjects: No more than a 30-day supply of study drug will be dispensed at a time.

Female Subjects:

* FCBP with regular cycles must agree to have pregnancy tests weekly for the first 28 days of study participation and then every 28 days while on study, at study discontinuation, and at day 28 following discontinuation from the study. If menstrual cycles are irregular, the pregnancy testing must occur weekly for the first 28 days and then every 14 days while on study, at study discontinuation, and at days 14 and 28 following discontinuation from the study.
* In addition to the required pregnancy testing, the Investigator must confirm with FCBP that she is continuing to use two reliable methods of birth control at each visit.
* Counseling about pregnancy precautions and the potential risks of fetal exposure must be conducted at a minimum of every 28 days. During counseling, subjects must be reminded to not share study drug and to not donate blood.
* Pregnancy testing and counseling must be performed if a subject misses her period or if her pregnancy test or her menstrual bleeding is abnormal. Study drug treatment must be discontinued during this evaluation.
* Females must agree to abstain from breastfeeding during study participation and for at least 28 days after discontinuation from the study.

Male Subjects:

* Counseling about the requirement for latex condom use during sexual contact with females of childbearing potential and the potential risks of fetal exposure must be conducted at a minimum of every 28 days. During counseling, subjects must be reminded to not share study drug and to not donate blood, sperm, or semen.
* If pregnancy or a positive pregnancy test does occur in a study subject or the partner of a male study subject during study participation, study drug must be immediately discontinued.

Exclusion Criteria:

* Subjects who are candidates for and willing to undergo an autologous stem cell transplant.
* Subjects who are post allogeneic stem cell transplant.
* All subjects with active central nervous system (CNS) lymphoma. Subjects with previous CNS lymphoma that have been treated with chemotherapy, radiotherapy or surgery who have remained asymptomatic for 90 days (3 months) and demonstrate, no CNS lymphoma, as shown by lumbar puncture, CT scan or MRI, are eligible. (If required, lumbar puncture, CT or MRI should be performed during screening process.) Subjects should not be receiving corticosteroids.
* Prior history of malignancies other than NHL (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless the subject has been free of the disease for > = 365 days (1 year).
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Known positive for HIV.
* Pregnant or lactating females.
* Concomitant Medications: Category I drugs that are generally accepted to have a risk of causing Torsades de Pointes including: (Patients must discontinue drug 7 days prior to starting dasatinib) quinidine, procainamide, disopyramide, amiodarone, sotalol, ibutilide, dofetilide, erythromycin, clarithromycin, chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide, cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone,halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine
* Concurrent medical condition which may increase the risk of toxicity, including:

  1. Pericardial or pleural effusion of any grade
  2. Clinically-significant coagulation or platelet function disorder (e.g. known von Willebrand's disease)
* History of significant bleeding disorder unrelated to cancer, including:

  1. Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease)
  2. Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)
  3. Ongoing or recent (< = 3 months) clinically significant gastrointestinal bleeding
* Cardiac symptoms within 6 months:

  1. Uncontrolled angina, congestive heart failure, or MI
  2. History of clinically significant ventricular arrythmias: fibrillation, Torsades de pointes, or tachycardia.
  3. Prolonged QTc interval on pre-entry electrocardiogram (> 450msec).
* Prior use of dasatinib.
* Use of any standard or experimental anti-cancer drug therapy within 28 days of the initiation (Day 1) of study drug therapy.
* Known active Hepatitis B or C.
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2011-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Elstrom, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Patients
Started | 2
Completed | 0
Not Completed | 2
Not completed — Death | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Response rate will be used as a measure of efficacy of dasatinib monotherapy in relapsed or refractory aggressive Diffuse Large B-Cell Lymphoma (DLBCL)
Time Frame: 2 years
Population: Data was not collected due to early termination of the study.
Arm/Group | All Patients
Number analyzed (Participants) | 0

2. Secondary Outcome: To Evaluate the Safety of Dasatinib Monotherapy as Treatment for Subjects With Relapsed or Refractory Aggressive DLBCL.
Time Frame: 2 years
Population: Data was not collected due to early termination of the study.
Arm/Group | All Patients
Number analyzed (Participants) | 0

3. Secondary Outcome: To Determine Potential Correlatives of Response.
Time Frame: 2 years
Population: Data was not collected due to early termination of the study.
Arm/Group | All Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Zero subjects at risk for "Other (Not Including Serious) Adverse Events" as subjects were not evaluated due to early study termination.
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=2)
Hypotension (Vascular disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No